CLINICAL TRIAL: NCT03080610
Title: Factors Influencing the Occurrence of Post Dural Puncture Headache in Patients Undergoing Cesarean Section After Epidural Blood Patch
Brief Title: The Occurrence of Post Dural Puncture Headache After Epidural Blood Patch
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Pattrapun Wongsripuemtet, Dr., Siriraj Hospital
Other Study IDs: Si 034/2012
Record Dates: First submitted 2017-03-03; First posted 2017-03-15 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Post-Dural Puncture Headache
Keywords: Post-Dural Puncture Headache [C10.228.140.546.699.124]; Blood Patch, Epidural [E02.319.267.530.580.300.145]
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal anesthesia is commonly used for cesarean section.However, the procedure is still have some adverse events such as high spinal block, nerve injuries or postdural puncture headache (PDPH).This is a potential complication of neuraxial anesthesia in clinical practice.

The investigators are curious regarding factors determining the incidence of postdural puncture headache in parturients undergoing cesarean section after epidural blood patch.

DETAILED DESCRIPTION:
Currently, spinal anesthesia is commonly used for cesarean section in many institutes, since it is a safe technique for both mother and child, with high satisfaction of obstetricians and their colleagues. Bloom, et al. claimed that there was 37,142 women underwent cesarean section in 2002 where 94% was under regional anesthesia, as 40% spinal, 42% epidural and 12% combined spinal and epidural anesthesia.

However, the procedure is inevitable to have some adverse events such as high spinal block, nerve injuries or postdural puncture headache (PDPH) . The PDPH is caused by accidental dura puncture resulting in continuous cerebrospinal fluid (CSF) leakage and gradual intracranial pressure reduction. This is a potential complication of neuraxial anesthesia in clinical practice. The needle characteristics as bevel orientation, stylet reinsertion, an approach, multiple insertion, and operator experience, patient age, history of previous PDPH, body mass index (BMI) > 35 are some responsible factors for the incidence. Chan et al. revealed that amongst 65,348 parturients, the occurence of PDPH was 1.1-1.9%, while Bloom et al. proposed his number as 0.4%. Interestingly, an obstetric meta-analysis showed an incidence of 1.5-11%, caused by spinal needle.

The PDPH is defined as a symptom of severe headache that appears within 7 days following a lumbar puncture. It may be accompanied by other manifestations such as tinnitus, hypoacusis, photophobia, nausea, or neck stiffness. Actually, it can resolve within 1 week or 48 hour after a treatment of blood patch. Other additional treatments include bed rest, analgesics, increase fluid intake, or caffeine containing beverages. In a severe case, a retractable pain might have a good response to intravenous caffeine and epidural blood patch (EBP). Though treatments of PDPH include both pharmacologic and non-pharmacologic regimens, Cochrane review concluded that the EBP was more effective than any other conservative treatments. As a result, the investigators are curious regarding factors determining the incidence of postdural puncture headache in parturients undergoing cesarean section after epidural blood patch.

ELIGIBILITY:
Inclusion Criteria:

* parturient after received spinal block for cesarean section who have post Dural puncture headache and received epidural blood patch in Siriraj hospital during 1 January 2006 to 30 December 2015

Exclusion Criteria:

* patient who diagnosed post Dural puncture headache from accidental Dural puncture from epidural needle or received combine spinal epidural anesthesia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: parturient after received spinal block for cesarean section who have post Dural puncture headache and received epidural blood patch.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
The Occurrence of Post Dural Puncture Headache after Epidural Blood Patch | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ladda Permpolprasert, B.N.S, Principal Investigator — Siriraj Hospital
Locations (2):
- Thailand (2):
  - Pattrapun Wongsripuemtet, Bangkok Noi, Bangkok
  - Pattrapun Wongsripuemtet, Bangkok

IPD SHARING:
Plan to Share IPD: No